CLINICAL TRIAL: NCT03151837
Title: A Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Hypoglycemic Efficacy of Greenyn Momordica Charantia Extracts in Diabetic Subjects
Brief Title: Hypoglycemic Efficacy of Greenyn Momordica Charantia Extracts in Diabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Nae-Cherng Yang, Associate Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS16148
Record Dates: First submitted 2017-04-26; First posted 2017-05-12 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Bitter melon(Momordica charantia); Insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Momordica charantia (Experimental): Subjects will take the capsule of Greenyn Momordica charantia extracts 600 mg/day orally for three months.
  Interventions: Dietary Supplement: Greenyn Momordica charantia extracts
- Placebo control (Placebo Comparator): Subjects will take the capsule of Placebo 600 mg/day orally for three months.
  Interventions: Dietary Supplement: Placebo control

INTERVENTIONS:
Dietary Supplement: Greenyn Momordica charantia extracts — Extracts from Momordica charantia containing Momordica charantia insulin receptor binding protein (mcIRBP)
  Arms: Momordica charantia
Dietary Supplement: Placebo control — Starch
  Arms: Placebo control

SUMMARY:
This is a randomized, double-blind, placebo-controlled, add-on clinical trial to evaluate the efficacy and safety of Momordica Charantia extracts taken orally for 3 months by subjects with type 2 diabetes. A total of 40 subjects who meet the inclusion criteria and give written consent will be randomly assigned to (A) Momordica charantia extracts group (600mg/day), or (B) Placebo group (Starch 600mg/day) with 20 subjects for each group. Major enrollment criteria include: (1)Subjects have confirmed type 2 diabetes and fail to reach the treatment goal (fasting glucose 140-270mg/dL and hemoglobin A1c (HbA1c) 7-10%) after stable use of 1-3 oral hypoglycemic drugs for 3 months; (2)Subjects have stable diabetes mellitus (DM) history with fasting glucose 140-270mg/dL and HbA1c 7-10% and refuse to use oral medications. Efficacy outcomes include the changes in fasting glucose, Hb1Ac, and insulin sensitivity, and safety assessments include liver and kidney function, and complains made by subjects after the initiation of the investigational products (IP).

DETAILED DESCRIPTION:
This study aims to investigate the hypoglycemic efficacy of oral Momordica Charantia extracts containing mcIRBP manufactured by Greenyn Biotechnology. The study objectives include:

1. To evaluate the changes in fasting glucose, hemoglobin A1c (Hb1Ac), glucose tolerance test, and insulin sensitivity after taking the investigational products (IP) orally for 3 months.
2. To evaluate the safety of the IP, including the liver and kidney function, and complains made by subjects after the initiation of the IP.

This is a randomized, double-blind, placebo-controlled, add-on clinical trial to evaluate the efficacy and safety of Momordica Charantia extracts taken orally for 3 months by subjects with type 2 diabetes. A total of 40 subjects who meet the enrollment criteria and give written consent will be randomly assigned to (A) Momordica charantia extracts group (600mg/day), or (B) Placebo group (Starch 600mg/day) with 20 subjects for each group. Subjects will take the IP for 12 weeks and the hypoglycemic medications taken by the subjects before enrollment will remain stable over the study period.

Study procedures for each visit:

Visit 1: Day 0

1. Obtain signed informed consent form
2. Assess vital signs and record concomitant medication
3. Lab tests: Fasting glucose, HbA1c, liver function, kidney function, hemoglobin (Hb)

Visit 2: <7 day from Visit 1

1. Confirm eligibility and randomization
2. Initiation of treatment
3. Lab tests: Fasting glucose, HbA1c, insulin, lipids, total protein, uric acid, oral glucose tolerance test (OGTT), ketone body
4. Measure height, weight, thigh circumference, waist and hip circumference
5. Record concomitant medication

Visit 3: 1 month after Visit 1

1. Measure vital signs
2. Lab tests: Fasting glucose, HbA1c, lipids, ketone body
3. IP Accountability and dispense IP
4. Records adverse events

Visit 4: 3 months after Visit 1

1. Lab tests: Fasting glucose, HbA1c, liver function, kidney function, Hb, insulin, lipids, total protein, uric acid, OGTT, ketone body
2. Measure vital signs, height, weight, thigh circumference, waist and hip circumference
3. IP Accountability and dispense IP
4. Records adverse events

Statistical Analysis All randomized subjects will be entered for efficacy analysis dataset, and subjects who receives at least one dose of IP will be included for safety analysis. Mean and standard deviation will be used for data presentation, and changes from baseline for all assessments will be plotted against time. Paired t test will be performed for the before and after treatment comparison within group, and 2-independent t test will be used to compare the changes from baseline between the two groups. All statistical analyses will be conducted by using SPSS v.18 (SPSS Inc., Chicago, IL, USA) and p<0.05 is considered to have statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 80 years of age
* Newly diagnosis with type 2 diabetes based on a fasting plasma glucose(FPG)>=126 mg/dL or 2-5 postprandial glucose levels during 75-g OGTT>=200 mg/dL
* The person who take 1-3 or more medicine to treat hyperglycemic but not very effective.(Fasting glucose:140-270mg/dL，HbA1c 7-10%)

Exclusion Criteria:

* Serum creatinine > 1.8mg/dL
* Serum ALT, AST, total bilirubin or alkaline phosphatase higher than 2.5 times of the upper normal range
* Anemia (Hb Male: < 11g/dL;Female: < 10g/dL)
* Pregnancy or Lactation
* Severe angina
* Moderate-severe heart failure with left ventricular hypertrophy
* BMI<18 or >38
* a body weight variation more than 10% during the screening period.
* Dietary habits change in one months or body weight change >10%
* Life expectancy is low than 6 months
* be allergy to bitter melon
* Severe long-term diabetic complications such as diabetic retinopathy,diabetic neuropathy,systemic orthostatic hypotension,urinary retention,foot ulcers or gastric stasis
* Acute disease
* Participation in another clinical trial within 30 days of screening

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-12-16 (Actual); Study Completion 2017-12-16 (Actual)

PRIMARY OUTCOMES:
Fasting glucose | from baseline at 3 month
  Fasting glucose in milligram per deciliter
Glycated hemoglobin | from baseline at 3 month
  Glycated hemoglobin in percentage
Fasting insulin | from baseline at 3 month
  Fasting insulin in milliunit per milliliter
Oral Glucose Tolerance Test | from baseline at 3 month
  Oral Glucose Tolerance Test in milligram per deciliter

SECONDARY OUTCOMES:
Total cholesterol | from baseline at 3 month
  Total cholesterol in milligram per deciliter
L.D.L.cholesterol | from baseline at 3 month
  L.D.L.cholesterol in milligram per deciliter
H.D.L.cholesterol | from baseline at 3 month
  H.D.L.cholesterol in milligram per deciliter
Body mass index(BMI) | from baseline at 3 month
  BMI in kg/m^2
Body fat | from baseline at 3 month
  Body fat in percentage
Waist circumference | from baseline at 3 month
  Waist circumference in centimeter
Hip circumference | from baseline at 3 month
  Hip circumference in centimeter
Upper arm circumference | from baseline at 3 month
  Upper arm circumference in centimeter
Ketone body | from baseline at 3 month
  Ketone body in positive or negative
total protein | from baseline at 3 month
  total protein in gram per deciliter
Blood pressure | from baseline at 3 month
  Blood pressure in millimeter of mercury
Aspartate Aminotransferase (AST) | from baseline at 3 month
  Aspartate Aminotransferase (AST) in IU per liter
Alanine Aminotransferase (ALT) | from baseline at 3 month
  Alanine Aminotransferase (ALT) in IU per liter
Creatinine | from baseline at 3 month
  Creatinine in milligram per deciliter
Blood urea nitrogen (BUN) | from baseline at 3 month
  BUN in milligram per deciliter
Uric Acid(UA) | from baseline at 3 month
  UA in milligram per deciliter
Hemoglobin(Hb) | from baseline at 3 month
  Hb in gram per deciliter

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Ning Huang, Ph.D., Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No